CLINICAL TRIAL: NCT00598923
Title: Preventing Epilepsy After Traumatic Brain Injury: A Pilot, Single-center Randomized Trial of Topiramate to Prevent Seizures After Moderate to Severe TBI
Brief Title: Preventing Epilepsy After Traumatic Brain Injury With Topiramate
Acronym: PEPTO
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: End of funding and low enrollment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR043514
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Traumatic Brain Injury; Epilepsy
Keywords: tbi; traumatic brain injury; epilepsy
MeSH Terms: conditions — Brain Injuries, Traumatic; Epilepsy | interventions — Topiramate; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Phenytoin 20mg/kg load, then Topiramate, 100 mg twice daily, starting at 24 hours post-TBI for 6 days.
  Interventions: Drug: topiramate
- 2 (Experimental): topiramate for 3 months after loading dose of phenytoin
  Interventions: Drug: topiramate
- 3 (Placebo Comparator): Phenytoin 20 mg/kg as loading dose than 300 mg/day for total of 7 days
  Interventions: Drug: phenytoin

INTERVENTIONS:
Drug: topiramate — 100 mg twice per day for 3 months
  Other Names: Topamax
  Arms: 2
Drug: topiramate — 100 twice per day for 6 days after loading dose of phenytoin
  Other Names: Topamax
  Arms: 1
Drug: phenytoin — loading dose of 20 mg/kg and then 300 mg/day for total of 7 days
  Other Names: Dilantin
  Arms: 3

SUMMARY:
Our hypothesis is that topiramate will reduce acute seizures after traumatic brain injury and will help prevent the development of epilepsy after traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) causes epilepsy in up to 30% of civilian and 50% of military head injuries, exacerbating chronic neurological disability. There is currently no method for preventing epilepsy after TBI. We hypothesize that the new antiepileptic drug, topiramate (TPM), will (1) reduce acute seizures and prevent the development of epilepsy following TBI and (2) improve neurological recovery. We propose to perform a pilot clinical trial to develop the necessary infrastructure for larger scale randomized clinical trials to test TPM, and, possibly, other new antiepileptic drugs with neuroprotective properties, for their ability to prevent epilepsy after TBI. Subjects with TBI will be randomized within 24 hours to one of three groups: 1) TPM for one week, 2) TPM for three months, or 3) phenytoin for one week. Subjects will be followed for two years for the development of seizures and for neurological outcome. Serial EEGs and MRIs will be performed to explore potential mechanisms for the development of epilepsy after TBI. These new tools for the clinical study of epilepsy prevention, and neuroprotection in general, will be developed that can be applied to a wide variety of studies and which will facilitate future research in this critical area.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe traumatic brain injury, defined as one or more of the following: penetrating head wound seizure within the first hour after injury intracerebral hematoma or cortical contusion subdural or epidural hematoma Glasgow Coma Score <= 12 or motor score 1-5 (if intubated). Patients who have been pharmacologically paralyzed will be evaluated after the paralytic has worn off or been pharmacologically reversed depressed skull fracture requirement for emergent neurosurgical procedure
2. Time since TBI less than 24 hours
3. Age greater than or equal to 18 years
4. Subject capable of giving informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf. -

Exclusion Criteria:

1. Known prior history of epilepsy or unprovoked seizures. Patients with a history of acute symptomatic seizures (e.g. febrile seizure, alcohol withdrawal seizure) will not be excluded
2. Administration of an antiepileptic drug before enrollment
3. History of allergy to topiramate or phenytoin
4. Pregnancy or breast-feeding. Women of childbearing potential must have a negative pregnancy test (urine pregnancy test or serum beta-HCG) before randomization
5. Compromised renal function with serum creatinine > 2
6. Severe concurrent illness with life expectancy <6 months
7. Treatment with another investigational agent for TBI
8. Unable to take medications orally and contraindication to placement of nasogastric tube.
9. Irreversibly fatal TBI

   1. All four findings: Glasgow Coma Score = 3, no pupillary reaction, age > 45 years, and severe coagulopathy OR
   2. Severe brainstem lesion on neuroimaging studies
10. Patients with a history of kidney stones or glaucoma.
11. Inability to maintain adequate fluid intake while taking topiramate.
12. Patients whose TBI is a result of self inflicted injury
13. Patient's who are currently using illicit drugs -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Early and late seizures after traumatic brain injury | 2 years
Adverse events | 2 years

SECONDARY OUTCOMES:
Functional recovery after traumatic brain injury | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Dichter, MD, PhD, Principal Investigator — University of Pennsylvania